CLINICAL TRIAL: NCT04719988
Title: Ezabenlimab (BI 754091) and mDCF (Docetaxel, Cisplatin and 5-fluorouracil) Followed by Chemoradiotherapy in Patients With Stage III Squamous Cell Anal Carcinoma. A Phase II Study
Brief Title: Anti-PD-1 and mDCF Followed by Chemoradiotherapy in Patients With Stage III Squamous Cell Anal Carcinoma.
Acronym: INTERACT-ION
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020/567
Record Dates: First submitted 2021-01-19; First posted 2021-01-22 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-11

CONDITIONS: Squamous Cell Carcinoma of the Anus Stage III
Keywords: immunotherapy; radiotherapy; chemotherapie; anal cancer
MeSH Terms: conditions — Anus Neoplasms | interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Induction treatment
  * Modified DCF: every 2 weeks for 8 cycles Docetaxel (40 mg/m², day 1), Cisplatin (40 mg/m², day 1) , 5-FU (1200 mg/m²/day for 2 days)
  * Ezabenlimab: 240 mg intravenous, every 3 weeks for 3 cycles
  In case of tumor response:
  * Two additional cycles of mDCF and one additional cycle of Ezabenlimab (Q3W).
  * Hypofractionated radiotherapy
  * Ezabenlimab: 240 mg intravenous, every 3 weeks for 7 cycles
  In absence of tumor response:
  o Chemoradiotherapy (Intensity-Modulated Radiation Therapy [IMRT]) treatment: Chemoradiotherapy using IMRT will begin 3-4 weeks following the last cycle of induction phase, in the absence of toxicities of grade 1 and/or management of toxicities. It will last 7 weeks and will consist of:
  • Standard dose of 45 Gy in 25 fractions over 5 weeks followed by a sequential boost of 14.4 Gy in 8 sessions,
  Concomitantly given with:
  * Capecitabine (825 mg/m²/orally twice daily) from Monday to Friday,
  * Mitomycin C (10 mg/m² Day 1)
  Interventions: Biological: Blood sample collection; Procedure: Biopsy

INTERVENTIONS:
Biological: Blood sample collection — A total of 9 EDTA (ethylenediaminetetraacetic acid) tubes will be collected at each time point to perform:
  PBMC collection: 6 EDTA tubes of 6 ml of peripheral blood mononuclear cell [PBMC] will be sent to the central laboratory (Biomonitoring Platform of Besançon, CHRU de Besançon located at Etablissement Français du Sang) at room temperature within 24 hours via an approved carrier for their processing, storage and immunomonitoring analysis. A sending sheet of the samples will be attached to each single sample.
  Plasma collection: One 6 ml EDTA tube should be frozen in each investigation center for plasma collection.
  Plasma for circulating tumoral DNA (ctDNA) collection: Two 4 ml EDTA tube should be frozen in each investigation center for ctDNA collection.
Procedure: Biopsy — A tumor biopsy will be performed at 2 months after enrollment.

SUMMARY:
Squamous cell carcinoma of the anus (SCCA) is a rare cancer, however its incidence is increasing worldwide. SCCA is mostly induced by human papillomavirus (HPV) infections (high-risk types such as HPV-16 and -18) and HPV-related oncoproteins (E6 and E7) are expressed in more than 90% of cases. T stage and N stage are recognized prognostic factors for local and/or distant recurrence in SCCA patients treated by CRT. In fact, ≥T3 or ≥N1 anal cancers are associated with as high as 50% disease recurrence rate at 2 years.

Since 1996 when concomitant radiotherapy and MMC (mytomicin C) and 5-FU-based chemotherapy demonstrated superiority to radiotherapy alone, no significant progress has been achieved in patients with locally advanced SCCA. Still, phase III study by James et al. reported in 2013 showed that prognosis of SCCA patients treated with this regimen can be improved probably due to a better tumor classification, more precise radiological methods, known as "Will Rogers phenomenon".

Based on the above, investigators have designed this phase II trial assessing the feasibility and efficacy of Ezabenlimab (BI 754091) and mDCF chemotherapy combination followed by:

* standard chemoradiotherapy in case of low response to induction treatment (<30% by RECIST criteria) or
* additional 2 cycles of mDCF and 1 cycle of Ezabenlimab (BI 754091) followed by hypofractionated radiotherapy in case of high response (≥ 30% by RECIST criteria)

in SCCA patients with high-risk locally advanced (stage III) disease.

In summary, the first innovative aspect of this research program is to provide a valuable proof of concept study evaluating the feasibility to combine radiotherapy, chemotherapies (docetaxel, cisplatin and 5-fluorouracil) and Ezabenlimab (BI 754091) in patients with stage III squamous cell anal carcinoma. INTERACT-ION study will provide evidence that Ezabenlimab (BI 754091) acts in synergy with mDCF to improve complete response rate, and both with hypofractionated radiotherapy to improve the disease-free survival enhancing TH1 and CD8 T cell immunity.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent,
* Age ≥18 years,
* Ability to comply with the study protocol in the Investigator's judgment,
* Performance status ECOG-WHO ≤ 1,
* Histologically proved squamous cell anal carcinoma,
* Locally advanced disease defined as:

  * Stage III (TxN1 or T4N0). Lymph node can be considered positive if one of the following criteria is satisfied:
  * Enlargement (largest short-axis diameter > 1 cm for mesorectal nodes, and > 1.5 cm for other nodes) OR,
  * Heterogeneity or necrosis OR,
  * Irregular contours OR,
  * Strong enhancement at magnetic resonance imaging (MRI) OR,
  * Positivity on positron emission tomography (PET) scan,
* Patient eligible to the mDCF regimen,
* Computed tomography (CT) scan performed within 30 days prior inclusion,
* MRI of pelvis performed within 30 days prior inclusion,
* PET scan performed within 30 days prior inclusion,
* Adequate hematologic and end-organ function: defined by the following laboratory test results obtained within 7 days prior to initiation of study treatment:

  * Absolute neutrophil count (ANC) ≥ 1.5 X 109/L (1500/µL),
  * Platelet count ≥ 100 X 109/L (100.000/µL) without transfusion,
  * Hemoglobin ≥ 90 g/L (9g/dL); previous transfusion is allowed,
  * Aspartate aminotransferase (AST), and alanine aminotransferase (ALT) ≤ 2.5 X upper limit of normal (ULN), (≤ 5 X upper limit of normal (ULN) if known liver metastases)
  * Serum bilirubin ≤ 2.5 X ULN (except patients with known Gilbert disease and serum bilirubin level ≤ 3 X ULN),
  * Creatinine clearance (CrCl) > 60 ml/min (by the Modification of Diet in Renal Disease [MDRD], Cockroft formula, or chronic kidney disease [CKD] formula]),
* Serum albumin ≥ 25 g/L (2.5 g/dL),
* For patients not receiving therapeutic anticoagulation: International normalized ratio (INR) or activated partial thromboplastin time (PTT) ≤ 1.5 X ULN,
* Patient affiliated to or beneficiary of French social security health insurance system.

Exclusion Criteria:

* Previously received chemotherapy or pelvic radiotherapy,
* Previously received anti-tumor immunotherapy (HPV vaccination is allowed),
* Metastatic disease,
* Diagnosis of additional malignancy within 3 years prior to the inclusion date with the exception of curatively treated basal cell carcinoma of the skin and/or curatively resected in situ cervical or breast cancer,
* Patient with any medical or psychiatric condition or disease, which would make the patient inappropriate for entry into this study,
* Current participation in a study of an investigational agent or in the period of exclusion,
* Pregnancy, breast-feeding or absence/refusal of adequate contraception for fertile patients during the period of treatment and for 6 months from the last treatment administration; men must refrain from donating sperm during this same period. In addition, men who are sexually active with woman of childbearing potential will be instructed to adhere to contraception for a period of 7 months after the last treatment administration,
* Female participants of childbearing potential and male participants with partners of childbearing potential must agree to use a highly effective method of birth control (i.e., pregnancy rate of less than 1% per year) during the study, A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus),
* Contraceptive methods that result in a low failure rate when used consistently and correctly include methods such as combined hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable), some intrauterine devices, intrauterine hormone-releasing stem, true sexual abstinence (when this is in line with the preferred and usual lifestyle of the participant), bilateral tubal occlusion, or a female partner who is not of childbearing potential or a male partner who has had a vasectomy. Women and female partners using hormonal contraceptive must also use a barrier method i.e. condom or occlusive cap (diaphragm or cervical/vault caps),
* Patient under guardianship, curatorship, or under the protection of justice
* Inadequate organ functions: uncontrolled cardiac condition, known cardiac failure, unstable coronaropathy, respiratory failure, and chronic obstructive pulmonary disease,
* Diabetes with vascular or neurovascular complications,
* Preexistent peripheral neuropathy or impaired audition,
* HIV positive with CD4 count under 400/mm3 (HIV test is mandatory before inclusion),
* Active hepatitis B virus (HBV) or active hepatitis C virus (HCV) infection (chronic or acute), defined as having a positive hepatitis B surface antigen (HBsAg) test at screening. Patients with a past or resolved HBV infection, defined as having a negative HBsAg test and a positive total HBV core antibody (HBcAb) test at screening, are eligible for the study. Active hepatitis C virus (HCV) infection, defined as having a positive HCV antibody test followed by a positive HCV RNA test at screening. The HCV RNA test will be performed only for patients who have a positive HCV antibody test,
* Active tuberculosis,
* Concomitant treatment with CYP3A4 inhibitor like ritonavir, indinavir, ketoconazole, etc,
* Known hypersensitivity or contraindication to any of the study chemotherapy drugs (taxanes, cisplatin, 5-FU, mitomycin, capecitabine) and dihydro pyrimidine dehydrogenase (DPD) deficit,
* Uncontrolled infection or another life-risk condition,
* Known hearing impairment that contraindicates cisplatin administration,
* Administration of a (attenuated) live vaccine within 28 days of planned start of study therapy of known need for this vaccine during treatment,
* Administration of prophylactic phenytoin,
* Inadequate laboratory values: MDRD CrCl < 60 ml/min, neutrophil count < 1500/mm3, platelets < 100.000/mm3, bilirubin 2.5 x ULN, AST/ALT 2.5 x ULN
* Previous major surgery (requiring general anesthesia) within 28 days of enrollment
* Any immunosuppressive therapy (i.e. corticosteroids > 10 mg of hydrocortisone or equivalent dose) within 14 days before the planned start of study therapy,
* Active autoimmune disease that has required a systemic treatment in past 2 years (i.e. corticosteroids or immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin) is allowed,
* Prior allogeneic bone marrow transplantation or prior solid organ transplantation,
* Known active central nervous system metastases and/or carcinomatous meningitis. Subject with previously treated brain metastases and with radiological and clinical stability are allowed,
* Previously received an anti-PD-1, anti-PD-L1, or anti-CTLA4 (Cytotoxic T-Lymphocyte Associated Protein 4) agent,
* Known hypersensitivity or allergy to Chinese hamster ovary cell products or any component of Ezabenlimab (BI 754091) formulation,
* History of colorectal inflammatory disease,
* History of idiopathic or secondary pulmonary fibrosis (History of radiation pneumonitis in the radiation field fibrosis is permitted), or evidence of active pneumonitis requiring a systemic treatment with 28 days before the planned start of study therapy
* History of severe hypersensitivity reactions to others mAbs
* History of Chronic colorectal inflammatory disease (Ulcerative colitis, Crohn's disease),
* History of connective disease,
* History of autoimmune diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2022-01-04 (Actual); Primary Completion 2024-11-21 (Actual); Study Completion 2026-07-05 (Estimated)

PRIMARY OUTCOMES:
Clinical complete response (cCR) at 10 months | 10 months
  The primary endpoint is the Clinical complete response (cCR) 10 months from the treatment initiation (the best time to evaluate the local response is 26 weeks from the commencement of standard CRT. In this protocol, with the neoadjuvant treatment, additional 14 weeks are necessary; ie 10 months). cCR rate at 10 months is defined as the number of patients alive without clinically detectable lesion and no residual disease by MRI or CT scan assessment at 10 months divided by the overall number of patients evaluable for cCR status at 10 months.
  A patient is evaluable for cCR status at 10 months if he dies during the 10 months of follow up or if he is alive with a RECIST evaluation available at 10 months.

CONTACTS AND LOCATIONS:
Overall Officials: Stefano KIM, Pr, Principal Investigator — CHU Besançon
Locations (10):
- France (10):
  - Centre Hospitalier Universitaire de Besançon, Besançon
  - Centre georges-François Leclerc, Dijon
  - Hôpital Franco-Britannique, Levallois-Perret
  - Centre Léon Bérard, Lyon
  - Hôpital Privé Jean Mermoz, Lyon
  - Hôpital Nord Franche-Comté, Montbéliard
  - Centre Antoine Lacassagne, Nice
  - Hôpital Saint Louis, Paris
  - CHU de Poitiers, Poitiers
  - CHU Robert Debré, Reims

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim S, Francois E, Andre T, Samalin E, Jary M, El Hajbi F, Baba-Hamed N, Pernot S, Kaminsky MC, Bouche O, Desrame J, Zoubir M, Ghiringhelli F, Parzy A, De La Fouchardiere C, Smith D, Deberne M, Spehner L, Badet N, Adotevi O, Anota A, Meurisse A, Vernerey D, Taieb J, Vendrely V, Buecher B, Borg C. Docetaxel, cisplatin, and fluorouracil chemotherapy for metastatic or unresectable locally recurrent anal squamous cell carcinoma (Epitopes-HPV02): a multicentre, single-arm, phase 2 study. Lancet Oncol. 2018 Aug;19(8):1094-1106. doi: 10.1016/S1470-2045(18)30321-8. Epub 2018 Jul 2. PMID 30042063
- [Background] Kim S, Meurisse A, Spehner L, Stouvenot M, Francois E, Buecher B, Andre T, Samalin E, Jary M, Nguyen T, El Hajbi F, Baba-Hamed N, Pernot S, Kaminsky MC, Bouche O, Desrame J, Zoubir M, Ghiringhelli F, Parzy A, de la Fouchardiere C, Boulbair F, Lakkis Z, Klajer E, Jacquin M, Taieb J, Vendrely V, Vernerey D, Borg C. Pooled analysis of 115 patients from updated data of Epitopes-HPV01 and Epitopes-HPV02 studies in first-line advanced anal squamous cell carcinoma. Ther Adv Med Oncol. 2020 Dec 4;12:1758835920975356. doi: 10.1177/1758835920975356. eCollection 2020. PMID 33329760
- [Derived] Kim S, Boustani J, Iseas S, Vernerey D, Evesque L, Quero L, Ghiringhelli F, Coutzac C, Bouche O, Chibaudel B, Vernet C, Vienot A, Tougeron D, Nguyen T, Rebucci-Peixoto M, Meurisse A, Chennoufi S, Maritaz C, Borg C; INTERACT-ION Study Team. Ezabenlimab and induction chemotherapy followed by adaptive chemoradiotherapy in patients with stage 3 squamous cell anal carcinoma (INTERACT-ION): an open-label, single-arm, phase 2 trial. Lancet Oncol. 2025 Dec;26(12):1626-1637. doi: 10.1016/S1470-2045(25)00605-9. Epub 2025 Nov 4. PMID 41202834
- [Derived] Kim S, Boustani J, Vernerey D, Vendrely V, Evesque L, Francois E, Quero L, Ghiringhelli F, de la Fouchardiere C, Dahan L, Bouche O, Chibaudel B, Hajbi FE, Vernet C, Rebucci-Peixoto M, Feuersinger A, Maritaz C, Borg C. Phase II INTERACT-ION study: ezabenlimab (BI 754091) and mDCF (docetaxel, cisplatin, and 5-fluorouracil) followed by chemoradiotherapy in patients with Stage III squamous cell anal carcinoma. Front Oncol. 2022 Aug 24;12:918499. doi: 10.3389/fonc.2022.918499. eCollection 2022. PMID 36119522